CLINICAL TRIAL: NCT03803020
Title: The Evaluation of Fractional Flow Reserve and D SPECT for the Intervention of Chronic Total Occlusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC12018X05
Record Dates: First submitted 2018-12-28; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; chronic total occlusion; fractional flow reserve; single-photon emission computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single coronary chronic total occlusion: symptomatic stable angina of single coronary chronic total occlusion without other coronary artery stenosis scheduled for elective PCI.
  fractional flow reserve and SPECT detection before and after intervention.
  Interventions: Other: fractional flow reserve and SPECT detection

INTERVENTIONS:
Other: fractional flow reserve and SPECT detection — fractional flow reserve and SPECT detection

SUMMARY:
Coronary chronic total occlusions (CTOs) are defined as an occluded coronary vessel with TIMI defined as an occluded coronary vessel with TIMI (Thrombolysis in Myocardial Infarction) grade flow 0 and an estimated duration of at least 3 months. They are frequently encountered in patients undergoing coronary angiography. The application of contemporary techniques and the use of advanced dedicated equipment lead to high procedural success and low adverse events rates in experienced centers. Fractional flow reserve (FFR) is a validated tool to assess physiological severity of coronary artery disease and have a prognostic role after percutaneous coronary intervention (PCI). SPECT (Single-Photon Emission Computed Tomography) is the golden standard for detection of myocardial ischemia. Recanalization of a CTO leads to a number of anatomical and pathophysiological changes to the coronary circulation. These include anatomical and functional collateral vessels regression and significant lumen enlargement because of recovery of blood flow and restoration of vasomotor tone. The effect of PCI on CTO is unknown. The aim of this study was to assess the functional result of CTO PCI by measuring FFR and D SPECT before and immediately post-CTO PCI and at short-term follow-up.

DETAILED DESCRIPTION:
Coronary chronic total occlusions (CTOs) are defined as an occluded coronary vessel with TIMI defined as an occluded coronary vessel with TIMI (Thrombolysis in Myocardial Infarction) grade flow 0 and an estimated duration of at least 3 months. They are frequently encountered in patients undergoing coronary angiography. The application of contemporary techniques and the use of advanced dedicated equipment lead to high procedural success and low adverse events rates in experienced centers. Fractional flow reserve (FFR) is a validated tool to assess physiological severity of coronary artery disease and have a prognostic role after percutaneous coronary intervention (PCI). SPECT (Single-Photon Emission Computed Tomography) is the golden standard for detection of myocardial ischemia. Recanalization of a CTO leads to a number of anatomical and pathophysiological changes to the coronary circulation. These include anatomical and functional collateral vessels regression and significant lumen enlargement because of recovery of blood flow and restoration of vasomotor tone. The effect of PCI on CTO is unknown. The aim of this study was to assess the functional result of CTO PCI by measuring FFR and D SPECT before and immediately post-CTO PCI and at short-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* single CTO lesions, or other stenosis have been PCI treated for more than one months
* the diameter of target vessel ≥2.5mm
* stable angina pectoris, or myocardial ischemia in the area of CTO lesions
* the patients agree to this research plan and sign the consent form, and complete the follow-up

Exclusion Criteria:

* Acute myocardial infarction in one month
* In addition to the area of CTO lesions, there are serious untreated coronary lesions
* bridge vascular CTO lesions
* untreated coronary artery or cardiac surgery due to interventional complications, or intraoperative death
* acute decompensated heart failure
* allergies to contrast or radionuclide tracers
* patients with planned pregnancies or lactation or 1 years after intervention
* malignant neoplasms or life expectancy of less than 1 years
* patients plan of surgery
* patients cannot tolerate double antiplatelet therapy for at least 12 months
* any condition that does not fit coronary intervention or is a drug-eluting stent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of single coronary chronic total occlusion
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
score of Seattle angina questionnaire | one year
  the result of Seattle angina questionnaire
socre of Self-Rating Anxiety Scale | one year
  result of socre of Self-Rating Anxiety Scale
socre of EuroQol five dimensions questionnaire | one year
  result of EuroQol five dimensions questionnaire
Composite of cardiac death, target vessel myocardial infarction and target lesion revascularization record in follow-up | one year
  Composite of cardiac death, target vessel myocardial infarction and target lesion revascularization record in follow-up
the success rate of Percutaneous Coronary Intervention | one year
  the success rate of Percutaneous Coronary Intervention

SECONDARY OUTCOMES:
rate of cardiac death rate | one year
  rate of cardiac death rate in one year recorded in follow-up
rate of target vessel revascularization rate | one year
  rate of target vessel revascularization rate in one year recorded in follow-up
rate of recurrent myocardial infarction rate | one year
  rate of recurrent myocardial infarction rate in one year recorded in follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jianying Ma, Doctor, Principal Investigator — Department of Cardiology, Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No